CLINICAL TRIAL: NCT03633175
Title: Efficacy of Prophylactic Vaginal Progesterone in Prevention of Preterm Delivery in Women With Placenta Previa
Brief Title: Progesterone in Patients With Placenta Previa
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohammed mahmoud samy, Lecturer in Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: progesterone
Record Dates: First submitted 2016-06-30; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal progesterone group (Active Comparator): Women will receive vaginal progesterone 400 mg [Prontogest® vaginal pessaries 400, Marcyrl, Cairo, Egypt], once at bed time starting from 26-28 weeks of gestation and till 36 weeks of gestation or delivery (which is closer).
  Interventions: Drug: Vaginal progesterone
- Control group (No Intervention): Women with gestational age from 26-28 weeks diagnosed with placenta previa who will not receive vaginal progesterone.

INTERVENTIONS:
Drug: Vaginal progesterone — 400 mg vaginal progesterone [Prontogest® vaginal pessaries 400, Marcyrl, Cairo, Egypt] will be given, once at bed time starting from 26-28 weeks of gestation till 36 weeks of gestation or delivery (which is closer).
  Other Names: Prontogest® suppositories
  Arms: Vaginal progesterone group

SUMMARY:
This study evaluates the efficacy of prophylactic vaginal progesterone administration in reducing of the episodes of antepartum hemorrhage and subsequent prevention of preterm delivery in women with placenta previa.

DETAILED DESCRIPTION:
Eligible women who consent to participate in the study are randomly allocated into one of the two study groups. Women who are allocated to the study group will receive vaginal progesterone 400 mg [Prontogest® vaginal pessaries 400, Marcyrl, Cairo, Egypt], once at bed time starting from 26-28 weeks of gestation and till 36 weeks of gestation or delivery (which is closer); while the other group will serve as controls. Patients will be followed up till delivery for the incidence in antepartum hemorrhagic episodes.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age 26-28 weeks of gestation.
2. Definite and reliable diagnosis of placenta previa (defined as presence of a placenta within 2 cm of the internal os), using a transvaginal ultrasound scan.

Exclusion Criteria:

1. Multiple pregnancy.
2. Women at high risk of preterm labor e.g. history of spontaneous preterm labor or preterm prelabor rupture of the membranes (PPROM).
3. Severe antepartum hemorrhage and/or hemodynamic instability that necessitates urgent intervention and delivery.
4. Women who have been maintained on progestin therapy since early pregnancy for whatever reason.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm delivery due to severe antepartum hemorrhage. | from 26 weeks till 37 weeks
  Number of patients who delivered before 37 weeks gestational age

SECONDARY OUTCOMES:
No. of episodes of antepartum hemorrhage. | from 26 weeks till 37 weeks
  Mean number of episodes of antepartum hemorrhage
Hospital admission for significant antepartum hemorrhage. | from 26 weeks till 37 weeks
  Number of patients requiring hospital admission for significant antepartum hemorrhage
Hospital admission for threatened preterm labor. | from 26 weeks till 37 weeks
  Number of patients requiring hospital admission for threatened preterm labor
Need for blood transfusion. | from 26 weeks till 37 weeks
  Number of patients requiring blood transfusion
Incidence of severe postpartum hemorrhage. | from 26 weeks till 37 weeks
  Number of patients who had severe postpartum hemorrhage
Incidence of Cesarean hysterectomy. | from 26 weeks till 37 weeks
  Number of patients who underwent cesarean hysterectomy
Patient compliance | from 26 weeks till 37 weeks
  measured as mean number of doses of vaginal progesterone missed per week
Patient satisfaction: Likert Scale | from 26 weeks till 37 weeks
  measured according to the 5-grade Likert scale: very unsatisfied, unsatisfied, indifferent, satisfied and very satisfied.
Neonatal Birth weight. | At birth
  measured in Kg
Need for NICU admission and its duration. | At birth
  Number of neonates needing NICU admission
Respiratory morbidity (transient tachypnea or respiratory distress syndrome). | At birth
  number of neonates with respiratory morbidities (transient tachypnea or respiratory distress syndrome).
Prematurity-related mortality. | 28 days postpartum
  Number of neonates dying due to prematurity-related cause

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samy, MD, Principal Investigator — M Samy
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: No